CLINICAL TRIAL: NCT04681248
Title: Expanded Access Use of DKN-01 for the Treatment of Advanced Solid Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DEK-DKK1-P206
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Neoplasm; Adenocarcinoma of the Gastroesophageal Junction; GastroEsophageal Cancer; Squamous Cell Carcinoma; Gastric Adenocarcinoma; Endometrial Cancer; Uterine Cancer; Ovarian Cancer; Carcinosarcoma; Gastric Cancer
Keywords: DKK1; DKN-01; epithelial histology; Wnt pathway; endometrial; uterine; ovarian; carcinosarcoma; gastric cancer; gastroesophageal junction
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Endometrial Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Carcinosarcoma; Stomach Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: DKN-01 — Administered by IV infusion

SUMMARY:
An Expanded Access Protocol for use of DKN-01 for the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a intermediate-size Expanded Access Protocol (EAP). Patients who were receiving DKN-01 in a parent study at the time of completion of the parent study, and are, in the opinion of the Investigator and Sponsor, suitable candidates for continued study drug treatment are eligible for participation in the current EAP. In this EAP, previously treated patients will receive DKN-01 at the same dose and schedule as at the time of completion of the parent study. Furthermore, patients who received DKN-01 in combination in the parent study will continue to receive the same combination agent at the same dose and schedule in the EAP.

DKN-01 naïve patients, with advanced solid tumors not eligible for enrollment to a DKN-01 clinical study but whom, in the opinion of the treating oncologist, would potentially receive benefit from treatment with DKN-01 while it is an investigational drug may be eligible for enrollment in this EAP. Eligible DKN-01 naïve patients with Wnt activating mutations will receive DKN-01 as monotherapy, administered intravenously on Day 1 of each 21-day cycle at a dose of 600 mg, with a loading dose of 600 mg of DKN-01 administered on Day 15 of Cycle 1 only.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed advanced solid tumors that are inoperable, locally advanced, metastatic, or recurrent, with no standard of care treatment options, and not eligible for enrollment to a DKN-01 clinical study, may be treated with DKN-01 in this study if in the opinion of the treating oncologist, would potentially receive benefit from treatment with DKN-01 while it is an investigational drug
* Prior documentation of a known Wnt activating mutation by a CLIA-accredited laboratory. Wnt activating mutations: CTNNB1, APC, AXIN1/2, RNF43, ZNRD3, RSPO2, RSPO3
* ECOG performance status (PS) of ≤ 2 (Medical Monitor's approval is needed for enrolling a patient with PS of 2).
* Laboratory values:

  1. Total bilirubin ≤ 2.0 times upper limit of normal (ULN). Total bilirubin must be < 3 X ULN for patients with Gilbert's syndrome.
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 X ULN (if liver metastases are present, then ≤ 5 X ULN is allowed).
  3. Serum creatinine ≤ 1.5 X ULN.
  4. Neutrophil absolute count ≥ 1,500/mm3 (≥1.5 X 109/L).
  5. Platelet count ≥ 75,000/mm3 (≥100 X 109/L).
  6. Hemoglobin ≥ 9g/dL (transfusion within 30 days of screening is permitted).

Exclusion Criteria:

* Major surgery within 4 weeks of first dose of study drug.
* Toxicities (as a result of prior anticancer therapy) that have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities).
* Any of the following cardiovascular risk factors:

  1. Pulmonary embolism within 28 days before first dose of study drug.
  2. Any history of acute myocardial infarction within 6 months before first dose of study drug.
  3. Uncontrolled hypertension that cannot be managed by standard anti-hypertension medications within 28 days before first dose of study drug.
* Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection within 14 days of first dose of study drug.
* Active brain metastases. Patients are eligible if brain metastases are adequately treated, and patients are neurologically stable for at least 2 weeks prior to enrolment without the use of corticosteroids or are on a stable or decreasing dose of ≤ 10mg daily prednisone (or equivalent).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - Cedars Sinai Medical Care Foundation, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin